CLINICAL TRIAL: NCT04406922
Title: The Impact of Circadian Rhythmicity in Cold-induced Thermogenesis in Lean and Obese Subjects
Brief Title: Circadian Rhythmicity in Cold-induced Thermogenesis
Acronym: COLDR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, mrboon, Principal Investigator, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: COLD_RHYTHM
Record Dates: First submitted 2020-01-21; First posted 2020-05-29 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Healthy; Obese; Glucose Intolerance
Keywords: lean; young; healthy; overweight; obese
MeSH Terms: conditions — Obesity; Glucose Intolerance; Overweight

STUDY DESIGN:
Intervention Model Description: The study design encompasses a single-arm randomized intervention study using cold exposure.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Cold exposure in the morning and evening.
  Interventions: Procedure: Personalized cooling protocol

INTERVENTIONS:
Procedure: Personalized cooling protocol — As an intervention, a personalized cooling protocol will be used in order to activate BAT and induce non-shivering thermogenesis. During the cooling procedure, subjects will be exposed to mild cold (approx. 14°C) for 150 min. Since the onset temperature of shivering shows a high interindividual variation, we will use a personal cooling protocol to ensure maximum non-shivering EE (and thus an equal maximum activation of BAT). The right temperature will be determined via a subjective method, e.g. to ask the subject if he or she experiences shivering. The time needed to achieve the right temperature is approximately 30-60 minutes. Then, the stable cooling period of 90 min is started. During this time the subject will be asked every 15 minutes whether he is experiencing shivering. If so, temperature will be increased with 2-3°C so that shivering just stops.

SUMMARY:
This study aims to investigate whether maximum cold-induced non-shivering thermogenesis (e.g. thermogenesis as a consequence of BAT activity) differs between morning and evening.

DETAILED DESCRIPTION:
Brown adipose tissue (BAT) recently emerged as a novel player in energy expenditure (EE) in humans as it combusts fatty acids and glucose towards heat. Human BAT can be activated by sympathetic stimulation resulting from cold exposure or treatment with sympathomimetic drugs. Short-term acclimation to mild cold was shown to reduce fat mass in obese subjects and decrease peripheral insulin resistance of patients with T2DM. Recently, in preclinical studies the investigators showed that BAT has a circadian rhythm. It is currently unknown whether this is also the case in humans. The investigators postulate that BAT activity should display a circadian rhythm that adapts to changes in circadian behavior, and may determine glucose/lipid levels throughout the day.

ELIGIBILITY:
Inclusion Criteria:

* Dutch white Caucasian males or females
* Age: 18-35 years
* Lean group: BMI ≥ 18 and ≤ 25 kg/m2
* Obese glucose tolerant group: BMI ≥ 30 and ≤ 42 kg/m2 and fasted plasma glucose levels < 5.5 and/or 2 h after OGTT ≤ 7.8 mM
* Obese impaired glucose tolerant group: BMI ≥ 30 and ≤ 42 kg/m2 and fasted plasma glucose levels ≥ 5.5 and/or 2 h after OGTT between 7.8 and 11.1 mM

Exclusion Criteria:

* Diabetes mellitus (determined on basis of fasting or OGTT defined by ADA criteria (30)
* Any other active endocrine disease (thyroid disease, any signs of Cushing's syndrome, adrenal disease and lipid-associated disorders such as familial hypercholesterolemia)
* Any chronic renal or hepatic disease
* Use of medication known to influence glucose and/or lipid metabolism or brown fat activity (e.g. beta blockers, antidepressants)
* Smoking
* Abuse of alcohol or other substances
* Pregnancy
* Participation in an intensive weight-loss program or vigorous exercise program during the last year before the start of the study
* Current participation in another research projects that may influence the current research project
* Clinically relevant abnormalities in clinical chemistry at screening (to be judged by the study physician)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Change in cold-induced non-shivering thermogenesis between morning and evening | Change in cold-induced non-shivering thermogenesis between morning (total duration of measurement 120 minutes) and evening (total duration of measurement 120 minutes). The time frame comprising both the morning and evening measurement will be 72 hours.
  Thermogenesis is estimated by the change in energy expenditure after cold exposure, measured by indirect calorimetry. This will be measured in the morning and in the evening.

SECONDARY OUTCOMES:
Change in glucose metabolism (mmol/L) | Change between morning and evening: measured at several timepoints during 3.5 hours. The time frame comprising both the morning and evening measurement will be 72 hours.
  Serum glucose (mmol/L) before and during cold exposure in the morning versus the evening.
Change in insulin (pmol/l) | Change between morning and evening: measured at several timepoints during 3.5 hours. The time frame comprising both the morning and evening measurement will be 72 hours.
  Serum insulin (pmol/l) before and during cold exposure in the morning versus in the evening.
Change in lipid metabolism (cholesterol) (mmol/L) | Change between morning and evening: measured at severaltime points during 3.5 hours. The time frame comprising both the morning and evening measurement will be 72 hours.
  Cholesterol (total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol) in serum (mmol/L). Before and during cold exposure in the morning and in the evening.
Change in lipid metabolism (triglycerides) (mmol/L) | Change between morning and evening: measured at severaltime points during 3.5 hours. The time frame comprising both the morning and evening measurement will be 72 hours.
  Triglycerides, glycerol and free fatty acids in serum (mmol/L). Before and during cold exposure in the morning and in the evening.
Change in markers for sympathetic output | Change between morning and evening: measured before and after cold exposure. The time frame comprising both the morning and evening measurement will be 72 hours.
  Norepinephrine, epinephrine (μM/ml)
Skin temperature | Change between morning and evening: measured every 60 seconds during cold exposure on both study days. The time frame comprising both the morning and evening measurement will be 72 hours.
  Wireless iButtons and infrared camera

CONTACTS AND LOCATIONS:
Overall Officials: Mariette R Boon, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sardjoe Mishre ASD, Straat ME, Martinez-Tellez B, Mendez Gutierrez A, Kooijman S, Boon MR, Dzyubachyk O, Webb A, Rensen PCN, Kan HE. The Infrared Thermography Toolbox: An Open-access Semi-automated Segmentation Tool for Extracting Skin Temperatures in the Thoracic Region including Supraclavicular Brown Adipose Tissue. J Med Syst. 2022 Nov 2;46(12):89. doi: 10.1007/s10916-022-01871-7. PMID 36319877
- [Derived] Straat ME, Martinez-Tellez B, Sardjoe Mishre A, Verkleij MMA, Kemmeren M, Pelsma ICM, Alcantara JMA, Mendez-Gutierrez A, Kooijman S, Boon MR, Rensen PCN. Cold-Induced Thermogenesis Shows a Diurnal Variation That Unfolds Differently in Males and Females. J Clin Endocrinol Metab. 2022 May 17;107(6):1626-1635. doi: 10.1210/clinem/dgac094. PMID 35176767